CLINICAL TRIAL: NCT02021786
Title: A Web- and Mobile Phone-based Intervention to Prevent Obesity in 4-year-olds (MINISTOP): a Population-based Randomized Controlled Trial
Brief Title: A web-and Mobile Phone-based Intervention in 4-year-olds: a Population-based Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Marie Löf, docent, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VF-2012-09062883
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobile phone based intervention (Experimental): The intervention in the present study is a web- and mobile phone based intervention aiming to develop healthy lifestyle behaviors regarding physical activity and dietary habits in 4-year-olds. The intervention will be delivered to the parents and it is available to the parents during six months.
  Interventions: Behavioral: Mobile phone based intervention
- Control (No Intervention): The control group receive a pamphlet on healthy eating and physical activity in pre-school children based on the existing guidelines. The information is similar to what parents receive from the Swedish child healthcare system

INTERVENTIONS:
Behavioral: Mobile phone based intervention — Parents in the intervention group receive a six month mHealth program (the MINISTOP app) based on social cognitive theory with strategies to change unhealthy diet and physical activity behaviors. The program includes information, advice, and strategies to change unhealty behaviours and the possibility to register the child's intake of fruits, vegetables, candy, sweetened beverages, moderate-to-vigorous physical activity, and sedentary time. Feedback is then provided on reported variables. In addition, the parents are able to ask questions through the app to a dietician and a psychologist.
  Arms: Mobile phone based intervention

SUMMARY:
This study aims to evaluate the effects of a mobile phone-based dietary and physical activity intervention on body fatness, dietary intake and physical activity of preschoolers

DETAILED DESCRIPTION:
Childhood overweight and obesity is an increasing health problem globally, and can be established as early as 2-5 years of age. Mobile phone based (mHealth) interventions have been successful for weight management in adults; however, their potential in young children is yet to be established. Therefore, the ultimate goal of MINISTOP (Mobile-based INtervention Intended to STop Obesity in Preschoolers) trial is to help parents of four year old children to achieve a healthy weight and body fat via a smartphone app (MINISTOP). More specifically this trial aims to reduce body fat (primary outcome), increase the intake of fruits, vegetables as well as decrease the intake of candy, and sweetened beverages, and increase the amount of time spent in moderate-to-vigorous physical activity and decrease sedentary behaviors (secondary outcomes) in healthy preschool aged Swedish children. If the MINISTOP app is effective, it has the potential to be incorporated into the child health care to aid in counteracting overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* parents having a four year old child and living in Östergötland; having the ability to have their child measured at baseline at 4.5 years ± 2 months of age
* at least one parent had to able to speak and read Swedish sufficiently well (i.e. be able to provide informed consent and understand the intervention content)

Exclusion Criteria:

* A child with a neurological or endocrine disease effecting weight
* A child with a parent suffering from a serious physical or psychological disease making the study too demanding for the family.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 315 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Body fat | At the end of the intervention and at a six month follow-up
  Fat mass index, FMI

SECONDARY OUTCOMES:
Diet and physical activity variables | At the end of the intervention and at a six month follow-up
  Fruit, vegetables, candy, sweetened beverages, sedentary time and physical activity

OTHER OUTCOMES:
Composite scores | At the end of the intervention and at a six month follow-up
  Two scores based on the primary and secondary outcomes. The first one contains all seven outcomes (body composition, dietary variables, and physical activity variables), while the second one only includes the six secondary outcomes (dietary and physical activity variables).

CONTACTS AND LOCATIONS:
Overall Officials: Marie Lof, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Biosciences and Nutrition, Karolinska Institute, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Delisle C, Sandin S, Forsum E, Henriksson H, Trolle-Lagerros Y, Larsson C, Maddison R, Ortega FB, Ruiz JR, Silfvernagel K, Timpka T, Lof M. A web- and mobile phone-based intervention to prevent obesity in 4-year-olds (MINISTOP): a population-based randomized controlled trial. BMC Public Health. 2015 Feb 7;15:95. doi: 10.1186/s12889-015-1444-8. PMID 25886009
- [Derived] Delisle Nystrom C, Sandin S, Henriksson P, Henriksson H, Maddison R, Lof M. A 12-month follow-up of a mobile-based (mHealth) obesity prevention intervention in pre-school children: the MINISTOP randomized controlled trial. BMC Public Health. 2018 May 24;18(1):658. doi: 10.1186/s12889-018-5569-4. PMID 29793467
- [Derived] Cadenas-Sanchez C, Henriksson P, Henriksson H, Delisle Nystrom C, Pomeroy J, Ruiz JR, Ortega FB, Lof M. Parental body mass index and its association with body composition, physical fitness and lifestyle factors in their 4-year-old children: results from the MINISTOP trial. Eur J Clin Nutr. 2017 Oct;71(10):1200-1205. doi: 10.1038/ejcn.2017.62. Epub 2017 May 3. PMID 28466851
- [Derived] Nystrom CD, Sandin S, Henriksson P, Henriksson H, Trolle-Lagerros Y, Larsson C, Maddison R, Ortega FB, Pomeroy J, Ruiz JR, Silfvernagel K, Timpka T, Lof M. Mobile-based intervention intended to stop obesity in preschool-aged children: the MINISTOP randomized controlled trial. Am J Clin Nutr. 2017 Jun;105(6):1327-1335. doi: 10.3945/ajcn.116.150995. Epub 2017 Apr 26. PMID 28446496